CLINICAL TRIAL: NCT05510232
Title: Influence of Virtual Reality Distraction on Pain and Satisfaction During Outpatient Pediatric Orthopedic Procedures: A Randomized Controlled Study
Brief Title: Virtual Reality Distraction During Outpatient Pediatric Orthopedic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0074
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Fractures, Bone; Deformity; Bone
MeSH Terms: conditions — Fractures, Bone; Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: Participants were randomized to each arm, with a target of 35 subjects in each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A treatment group that will watch a non-VR video via an iPad (Experimental): Demographic appropriate screening for inclusion ( including age and available past medical history)
  Patient consent (before randomization),
  iPad administration (description below),
  cast sawing,
  physical examination (before and after procedure),
  pulse oximetry application (HR measured 3 minutes pre-procedure and throughout entire procedure),
  NRS VAS pain administration (3 minutes pre-procedure and immediately post-procedure) in patients over 8 years(Will mark on scale),
  VAS Faces pain administration (3 minutes pre-procedure and immediately post-procedure) in patients under 8 years (Will point to face),
  NRS VAS anxiety administration (3 minutes pre-procedure and immediately post-procedure)(Will mark on scale),
  VAS Faces anxiety scale administration in patients under 8 years(Will point to face),
  Patient/parent satisfaction administration (post-procedure).
  Interventions: Device: A treatment group that will watch a non-VR video via an iPad
- A treatment group that will have headset on and will watch a VR video (Experimental): Demographic appropriate screening for inclusion ( including age and available past medical history)
  Patient consent (before randomization),
  Video administration via headset(description below),
  Cast sawing,
  Physical examination (before and after procedure),
  Pulse oximetry application (HR measured 3 minutes pre-procedure and throughout entire procedure),
  NRS VAS pain administration (3 minutes pre-procedure and immediately post-procedure) in patients over 8 years(Will mark on scale),
  VAS Faces pain administration (3 minutes pre-procedure and immediately post-procedure)in patients under 8 years(Will point to face),
  NRS VAS anxiety administration (3 minutes pre-procedure and immediately post-procedure)(Will mark on scale),
  VAS Faces anxiety administration (3 minutes pre-procedure and immediately post-procedure) in patients under 8 years (Will point to face),
  Patient/parent satisfaction administration (post-procedure).
  Interventions: Device: A treatment group that will have headset on and will watch a non-VR video
- A treatment group that will be immersed in the VR game (Bear Blast) via the headset. (Experimental): Demographic appropriate screening for inclusion ( including age and available past medical history)
  Patient consent (before randomization)
  VR assembly and administration (description below)
  Cast sawing,
  physical examination (before and after procedure) ,
  pulse oximetry application (HR measured 3 minutes pre-procedure and throughout entire procedure),
  NRS VAS pain administration (3 minutes pre-procedure and immediately post-procedure) in patients over 8,-(Will mark on scale)
  VAS Faces pain administration (3 minutes pre-procedure and immediately post-procedure) in patients under 8 years(Will point to face),
  NRS VAS anxiety administration (3 minutes pre-procedure and immediately post-procedure)(Will mark on scale),
  VAS Faces anxiety scale administration (3 minutes pre-procedure and immediately post-procedure) in patients under 8 years(Will point to face),
  Patient/parent satisfaction administration (post-procedure).
  Interventions: Device: A treatment group that will be immersed in the VR game (Bear Blast) via the headset.

INTERVENTIONS:
Device: A treatment group that will watch a non-VR video via an iPad — The iPad is a tablet computer first offered by Apple in 2010.The device resembles a much larger version of Apple's iPhone or its iPod Touch, and is about the same size as a magazine.The iPad uses the same operating system as the Apple iPhone, and uses very similar hardware. iPad will be used to deliver non VR video to patients.
  A standardized age appropriate video will be used for patients between ages 4-9 and a different standardized age appropriate video for patients ages 10-14. The selected videos will be the same for both the cast and suture/pin removal groups.
  Arms: A treatment group that will watch a non-VR video via an iPad
Device: A treatment group that will have headset on and will watch a non-VR video — Oculus headset will deliver VR video to patients. Headset will be administered before intervention and removed at the completion of the intervention unless patient requests otherwise. Patients visual field will not change with head motion and will remain static throughout cast removal or pin/suture removal.
  A standardized age appropriate video will be used for patients between ages 4-14. The selected videos will be the same for both the cast and suture/pin removal groups.
  Arms: A treatment group that will have headset on and will watch a VR video
Device: A treatment group that will be immersed in the VR game (Bear Blast) via the headset. — VR using the Oculus headset will deliver VR images and sound. Patients will watch a 15-minute VR experience called Bear Blast. Bear Blast is an immersive, 360-degree, game experience that takes place in a fantasy world where the user attempts to shoot balls at a wide range of moving objects by gently maneuvering his or her head toward the targets. Bear Blast is a nonviolent and noncompetitive game that incorporates motivational music and features positively reinforcing sounds, animation, and direct messages to patients. Bear Blast will be used as the standardized game for all patients in the VR group of both study arms. The VR Oculus headset can be controlled entirely via head motion and does not involve the use of patients extremities.
  Arms: A treatment group that will be immersed in the VR game (Bear Blast) via the headset.

SUMMARY:
Virtual Reality(VR) has had promising applications in science and medicine, including intervention delivery. The use of VR interventions has been studied in a wide range of medical conditions, including anxiety, phobias, obesity, chronic pain, and eating disorders. VR based simulation in pediatrics has grown rapidly in recent years and is expected to continue to grow. VR technology has become increasingly affordable, flexible, and portable, enabling its use in a broad range of environments including the outpatient clinical setting. Additionally, children are believed to have an inclination toward games of "pretend" or alternate realities further indicating the potential of this technology. While immersed in a game, they often become deeply absorbed and able to ignore aversive stimuli. VR is an engaging intervention that may help to detract from pain and anxiety for children undergoing painful procedures. Heart rate has been used as a means to objectively quantify the physiologic response to pain and anxiety.

The purpose of the study is to conduct a randomized controlled study that assess the utility of Virtual Reality simulations compared to non immersive visual distraction in pediatric patients undergoing outpatient procedures including cast removal and surgical suture/pins removal. Primary outcomes will include changes in patient heart rate (an age-validated surrogate for pain and anxiety) and patient-reported changes in anxiety and pain. Secondary outcomes will include patient/parent-reported satisfaction.

DETAILED DESCRIPTION:
Cast, pin and suture removal are involved in post-procedural pediatric orthopedic care. Although viewed as straightforward and routine parts of outpatient management, they may be viewed as painful, and serve as a source of anxiety for patients. A randomized control trial by Lim et al investigated the potential for analgesia to decrease the pain perception experienced during pin removal. The authors failed to identify a statistically significant decrease in heart rate and pain score during pin removal with ibuprofen or acetaminophen treatment compared to placebo. The failure of analgesia to produce a significant change in pain perception and heart rate of pediatric patients may indicate that there is a psychological component of this pain and anxiety that is poorly understood and can potentially be altered.

The absence of a standard intervention to decrease the morbidity associated with pin, suture and cast removal warrants further investigation into alternate interventions that could be helpful. The well described capacity of Virtual Reality to modulate subjective experiences especially in the pediatric population makes it a compelling intervention in the acute clinical setting. To date, no studies have explored the utilization of VR as a means of decreasing the morbidity associated with outpatient orthopedic interventions such as pin, suture and cast removal has currently not been investigated.

Virtual reality(VR) has garnered interest in a number of medical domains and clinical settings. VR technology has also proven efficacy in the domain of pain management and neurorehabilitation. VR has also found application in the pediatric population. VR has also been found useful as a distraction technique in acute care pediatric procedures such as phlebotomy. Schmitt et al investigated the use of VR in dressing changes for pediatric patients who had sustained burn wounds. Their work demonstrated a pain score reduction of 27-44% in pediatric patients who participated in the virtual reality gaming environment while undergoing dressing changes.

Casts, sutures and pins are often utilized as primary or adjunct interventions and removed weeks after the intended healing goals are met. In clinical practice, pain and anxiety are often experienced by pediatric patients during outpatient suture, pin or cast removal. Heart rate has been used extensively in the objective quantification of the pain response in the pediatric population. To capture the subjective sensation of pain and anxiety, the Visual Analog Scale (VAS) is pain scale is commonly utilized. Lim et al conducted a randomized control trials looking at the potential for analgesia to decrease the pain perception experienced during pin removal. The authors failed to identify a statistically significant decrease in the pain score with ibuprofen or acetaminophen treatment vs. placebo treatment. The failure of analgesia to produce a significant change in pain perception and heart rate of pediatric patients may indicate that the dissatisfaction related to the experience of pin or suture removal may not entirely be related to the parameters investigated by the study.

Similarly, casting is a routine procedure used for the treatment fractures in the pediatric population. Casting can be used to immobilize non-displaced fractures and stabilize the reduction of displaced fractures. Cast removal in the pediatric population can also be a challenge for patients, parents and providers. The fear and anxiety experienced by pediatric patients during cast removal can adversely impact the clinical encounter. Noise reduction and music therapy have been used for cast removal in pediatric patients have shown promise in smaller RCT's that have reported reduced heart rates during intervention delivery. Studies showing the efficacy of distraction techniques in decreasing patient pain and anxiety question if more immersive distractions, such virtual reality gaming, could have the potential to positively influence the the outpatient pediatric orthopedic experience.

The purpose of the study is to assess the utility of Virtual Reality simulations in pediatric patients undergoing outpatient interventions including cast and surgical suture/pins removal. Primary outcomes will include changes in patient heart rate and patient-reported changes in anxiety and pain with virtual reality assisted treatment. Secondary outcomes will include patient reported satisfaction and procedure disturbance count as quantified by the number of times a patient looks over at the site of intervention.

ELIGIBILITY:
Inclusion Criteria:

-All patients pediatric patients undergoing cast, pin and suture removal between the ages of 4 -14 years

Exclusion Criteria:

* History of epilepsy and seizures
* Anxiety disorders documented
* Unable to understand/follow VR directions
* History of vertigo and/or dizziness
* History of chronic pain
* Non-English speakers

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 226 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Fabricant, MD, MPH, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some participants did not tolerate the distraction method (e.g. removed virtual reality headset) or removed the heart rate monitor.
Groups:
- A Treatment Group That Will Watch a Non-VR Video Via an iPad: A treatment group that will watch a non-VR video via an iPad: The iPad is a tablet computer first offered by Apple in 2010.The device resembles a much larger version of Apple's iPhone or its iPod Touch, and is about the same size as a magazine. The iPad uses the same operating system as the Apple iPhone, and uses very similar hardware. iPad will be used to deliver non VR video to patients.
  A standardized age appropriate video will be used for patients between ages 414. The selected videos will be the same for both the cast and suture/pin removal groups.
- A Treatment Group That Will Have Headset on and Will Watch a VR Video: A treatment group that will have headset on and will watch a VR video: Oculus headset will deliver non VR video to patients. Headset will be administered before intervention and removed at the completion of the intervention unless patient requests otherwise. Patients visual field will not change with head motion and will remain static throughout cast removal or pin/suture removal.
  A standardized age appropriate video will be used for patients between ages 414. The selected videos will be the same for both the cast and suture/pin removal groups.
Period: Overall Study
Arm/Group | A Treatment Group That Will Watch a Non-VR Video Via an iPad | A Treatment Group That Will Have Headset on and Will Watch a VR Video | A Treatment Group That Will be Immersed in the VR Game (Bear Blast) Via the Headset.
Started | 76 | 80 | 70
Completed | 74 | 73 | 64
Not Completed | 2 | 7 | 6
Not completed — Withdrawal by Subject | 2 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- A Treatment Group That Will Watch a Non-VR Video Via an iPad: A treatment group that will watch a non-VR video via an iPad: The iPad is a tablet computer first offered by Apple in 2010.The device resembles a much larger version of Apple's iPhone or its iPod Touch, and is about the same size as a magazine. The iPad uses the same operating system as the Apple iPhone, and uses very similar hardware. iPad will be used to deliver non VR video to patients.
  A standardized age appropriate video will be used for patients between ages 4-14. The selected videos will be the same for both the cast and suture/pin removal groups.
- A Treatment Group That Will Have Headset on and Will Watch a VR Video: A treatment group that will have headset on and will watch a VR video: Oculus headset will deliver VR video to patients. Headset will be administered before intervention and removed at the completion of the intervention unless patient requests otherwise. Patients visual field will not change with head motion and will remain static throughout cast removal or pin/suture removal.
  A standardized age appropriate video will be used for patients between ages 4-14. The selected videos will be the same for both the cast and suture/pin removal groups.
- A Treatment Group That Will be Immersed in the VR Game (Bear Blast) Via the Headset.: A treatment group that will be immersed in the VR game (Bear Blast) via the headset.: VR using the Oculus headset will deliver VR images and sound. Patients will watch a 15-minute VR experience called Bear Blast. Bear Blast is an immersive, 360-degree, game experience that takes place in a fantasy world where the user attempts to shoot balls at a wide range of moving objects by gently maneuvering his or her head toward the targets. Bear Blast is a nonviolent and noncompetitive game that incorporates motivational music and features positively reinforcing sounds, animation, and direct messages to patients. Bear Blast will be used as the standardized game for all patients in the VR group of both study arms. The VR Oculus headset can be controlled entirely via head motion and does not involve the use of patients extremities. iPad will be set up and held for patients in the iPad group.
- Total: Total of all reporting groups
Arm/Group | A Treatment Group That Will Watch a Non-VR Video Via an iPad | A Treatment Group That Will Have Headset on and Will Watch a VR Video | A Treatment Group That Will be Immersed in the VR Game (Bear Blast) Via the Headset. | Total
Number analyzed (Participants) | 76 | 80 | 70 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 76 | 80 | 70 | 226
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9 (3) | 9 (3) | 9 (3) | 9 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 43 | 29 | 110
  Male | 38 | 37 | 41 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 6 | 21
  Not Hispanic or Latino | 60 | 67 | 55 | 182
  Unknown or Not Reported | 7 | 7 | 9 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 11 | 7 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 7 | 17
  White | 46 | 51 | 35 | 132
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 22 | 13 | 21 | 56
Region of Enrollment [Number; unit: participants]
  United States | 76 | 80 | 70 | 226

OUTCOME MEASURES:

1. Primary Outcome: Absolute Difference in HR as Measured 3 Minutes Prior to Procedure and Maximum as Measured During Through 1 Minute After Procedure.
Description: Pulse oximetry application
Time Frame: 3 minutes pre-procedure until 1 minute post-procedure, up to 20 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- A Treatment Group That Will Have Headset on and Will Watch a Non-VR Video: A treatment group that will have headset on and will watch a VR video: Oculus headset will deliver VR video to patients. Headset will be administered before intervention and removed at the completion of the intervention unless patient requests otherwise. Patients visual field will not change with head motion and will remain static throughout cast removal or pin/suture removal.
  A standardized age appropriate video will be used for patients between ages 4-14. The selected videos will be the same for both the cast and suture/pin removal groups.
- A Treatment Group That Will be Immersed in the VR Game (Bear Blast) Via the Headset.: A treatment group that will be immersed in the VR game (Bear Blast) via the headset.: VR using the Oculus headset fitted with a Samsung Galaxy S7 phone will deliver VR images and sound. Patients will watch a 15-minute VR experience called Bear Blast. Bear Blast is an immersive, 360-degree, game experience that takes place in a fantasy world where the user attempts to shoot balls at a wide range of moving objects by gently maneuvering his or her head toward the targets. Bear Blast is a nonviolent and noncompetitive game that incorporates motivational music and features positively reinforcing sounds, animation, and direct messages to patients. Bear Blast will be used as the standardized game for all patients in the VR group of both study arms. The VR Oculus headset can be controlled entirely via head motion and does not involve the use of patients extremities. iPad will be set up and held for patients in the iPad group.
Arm/Group | A Treatment Group That Will Watch a Non-VR Video Via an iPad | A Treatment Group That Will Have Headset on and Will Watch a Non-VR Video | A Treatment Group That Will be Immersed in the VR Game (Bear Blast) Via the Headset.
Number analyzed (Participants) | 74 | 73 | 64
beats per minute | 20 (16) | 20 (16) | 21 (16)

2. Secondary Outcome: Difference in Visual Analogue Scale (VAS) Pain Score as Measured 3 Minutes Before and Immediately After Intervention
Description: Difference in VAS pain score as measured 3 minutes before and immediately after intervention. This score is measured on a scale from 0-10, with 10 meaning the worst pain.
Time Frame: 3 minutes before and immediately after intervention
Reporting Status: Not Posted

3. Secondary Outcome: Difference in Visual Analogue Scale (VAS) Anxiety Score as Measured 3 Minutes Before and Immediately After Intervention
Description: Difference in VAS anxiety score as measured 3 minutes before and immediately after intervention. This score is measured on a scale from 0-10, with 10 meaning the worst anxiety.
Time Frame: 3 minutes before and immediately after intervention
Reporting Status: Not Posted

4. Secondary Outcome: Parent/Guardian Post-procedure Satisfaction Questionnaire Response
Description: Parent/guardian satisfaction is measured by a question asking the parent/guardian's satisfaction with the entire procedure on a scale from 1-10, where 10 is the most satisfied.
Time Frame: Immediately after intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During the procedure, an average of 30 minutes.
Arm/Group | A Treatment Group That Will Watch a Non-VR Video Via an iPad | A Treatment Group That Will Have Headset on and Will Watch a VR Video | A Treatment Group That Will be Immersed in the VR Game (Bear Blast) Via the Headset.
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/80 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/80 | 0/70
Other Adverse Events (participants affected / at risk) | 0/76 | 0/80 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT05510232/Prot_SAP_000.pdf